CLINICAL TRIAL: NCT07381075
Title: A Randomized, Non-comparative, Multicenter Phase II Clinical Trial of Becotatug Vedotin Combined With or Without Immune Checkpoint Inhibitors (Penpulimab/Ivonescimab) in the Neoadjuvant Treatment of Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: A Phase II Clinical Trial of Anti-EGFR Antibody-drug Conjugate (ADC) Combined With or Without Immune Checkpoint Inhibitors in the Neoadjuvant Treatment of Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lei Liu, professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRG003-IIT-2026
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Locally advanced head and neck squamous cell carcinoma; Neoadjuvant therapy; Antibody drug conjugate; Immunotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — penpulimab

STUDY DESIGN:
Intervention Model Description: A Randomized, Non-comparative, Multicenter Phase II Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Becotatug Vedotin (Experimental): Subjects receive 3 cycles of Becotatug Vedotin (2.3mg/kg, ivgtt, every 3 weeks, D1). Dose adjustments are allowed based on toxicity. Surgery will be performed within 2 to 4 weeks after the completion of neoadjuvant therapy, with subsequent adjuvant radiotherapy or chemoradiotherapy based on risk factors after surgery.
  Interventions: Drug: Becotatug Vedotin
- Becotatug Vedotin Combined with Penpulimab (Experimental): Subjects receive 3 cycles of Becotatug Vedotin (2.3mg/kg, ivgtt, every 3 weeks, D1) and 3 cycles of Penpulimab (200mg, ivgtt, every 3 weeks, D1). Surgery will be performed within 2 to 4 weeks after the completion of neoadjuvant therapy, with subsequent adjuvant radiotherapy or chemoradiotherapy based on risk factors after surgery. Subjects will receive Penpulimab treatment for 14 cycles following the completion of radiotherapy.
  Interventions: Drug: Becotatug Vedotin Combined with Penpulimab
- Becotatug Vedotin Combined with Ivonescimab (Experimental): Subjects received 3 cycles of Becotatug Vedotin (2.3mg/kg, ivgtt, every 3 weeks, D1) and 3 cycles of Ivonescimab (10mg/kg, ivgtt, every 3 weeks, D1). Dose adjustments are allowed based on toxicity. Surgery will be performed within 2 to 4 weeks after the completion of neoadjuvant therapy, with subsequent adjuvant radiotherapy or chemoradiotherapy based on risk factors after surgery. Subjects will receive Ivonescimab treatment for 14 cycles following the completion of radiotherapy.
  Interventions: Drug: Becotatug Vedotin Combined with Ivonescimab

INTERVENTIONS:
Drug: Becotatug Vedotin — Subjects receive 3 cycles of Becotatug Vedotin (2.3mg/kg, ivgtt, every 3 weeks, D1).
  Arms: Becotatug Vedotin
Drug: Becotatug Vedotin Combined with Penpulimab — Subjects receive 3 cycles of Becotatug Vedotin (2.3mg/kg, ivgtt, every 3 weeks, D1) and 3 cycles of Penpulimab (200mg, ivgtt, every 3 weeks, D1).
  Arms: Becotatug Vedotin Combined with Penpulimab
Drug: Becotatug Vedotin Combined with Ivonescimab — Subjects received 3 cycles of Becotatug Vedotin (2.3mg/kg, ivgtt, every 3 weeks, D1) and 3 cycles of Ivonescimab (10mg/kg, ivgtt, every 3 weeks, D1).
  Arms: Becotatug Vedotin Combined with Ivonescimab

SUMMARY:
A Randomized, Non-comparative, Multicenter Phase II Clinical Trial of Becotatug Vedotin Combined with or without Immune Checkpoint Inhibitors (Penpulimab/Ivonescimab) in the Neoadjuvant Treatment of Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma (LAHNSCC). This proposed study will evaluate the efficacy and safety of preoperative administration of Becotatug Vedotin Combined with or without Immune Checkpoint Inhibitors (Penpulimab/Ivonescimab) in LAHNSCC who are eligible for resection.

DETAILED DESCRIPTION:
In this study, eligible patients will be randomized in a 1:1:1 ratio to either the Becotatug Vedotin treatment group (Cohort 1), or the Becotatug Vedotin combined with Penpulimab treatment group (Cohort 2), or the Becotatug Vedotin combined with Ivonescimab treatment group (Cohort 3). Pathological response rate will be the primary outcome measures. Adverse events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 70 years old, gender not restricted;
2. Histopathologically diagnosed as squamous cell carcinoma of the head and neck (including oral cancer, laryngeal cancer, hypopharyngeal cancer, and oropharyngeal cancer, etc.);
3. Patients with resectable locally advanced head and neck squamous cell carcinoma (LA-HNSCC);
4. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1;
5. Have not received any treatment for head and neck squamous cell carcinoma before, including drug treatment, radiotherapy, surgical treatment, etc.;
6. No distant metastasis;
7. The patient has the intention for radical treatment;
8. Good hematopoietic function (total white blood cell count ≥ 3.0×109 /L, absolute lymphocyte count ≥ 0.8×109/L, absolute neutrophil count ≥ 1.5×109/L, platelet count ≥ 100×109 /L, hemoglobin ≥ 90g/L) and no blood transfusion or biological response modifiers (such as granulocyte growth factors, erythropoietin growth factors, etc.) treatment within 14 days before the first administration;
9. Good liver function (total bilirubin (TBIL) ≤ 1.5×ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤ 2.5×ULN; serum albumin ≥ 28 g/L);
10. Good renal function (serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance rate ≥ 50 mL/min (Cockcroft-Gault formula), urine protein less than 2+, or 24-hour urine protein quantification < 1g);
11. Good cardiac function, that is, normal electrocardiogram or abnormal without clinical significance, and echocardiography shows left ventricular ejection fraction (left ventricular ejection fraction, LVEF) ≥ 50%;
12. Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN, if the subject is receiving anticoagulation treatment, as long as the PT is within the range of the anticoagulant drug plan, it is acceptable;
13. During the screening period, blood pressure is well controlled (defined as systolic blood pressure ≤ 150 mmHg and diastolic blood pressure ≤ 90 mmHg), and there is no change in antihypertensive treatment within 1 week before the first administration of the study drug;
14. Patients with HBV infection who can detect HBV deoxyribonucleic acid (DNA) levels (≥ 10IU/mL or above the detection limit) must receive antiviral treatment before randomization according to the clinical institution practice to ensure adequate viral suppression. Patients must maintain antiviral treatment during the study and within 6 months after the last study treatment administration. Patients with positive Anti-HBc detection but no HBV DNA ( < 10IU/mL or below the detection limit) do not require antiviral treatment, unless HBV DNA exceeds 10IU/mL or above the detection limit during the treatment period;
15. Male patients with fertility and women of childbearing age who are willing to take effective contraceptive measures from signing the informed consent form to the last administration of the study drug within 6 months; women of childbearing age include pre-menopausal women and post-menopausal women within 1 year. The blood pregnancy test result of women of childbearing age within ≤ 7 days before the first administration of the study drug must be negative;
16. The subject voluntarily joins the study, signs the informed consent form, has good compliance, and cooperates with follow-up.

Exclusion Criteria:

1. Has received any form of anti-tumor treatment before;
2. Patients with allergic constitution and congenital immune deficiency;
3. Has undergone organ transplantation before;
4. Has a history of severe bleeding tendency or coagulation dysfunction; had significant clinical bleeding symptoms within 1 month before the study treatment, including but not limited to gastrointestinal bleeding and hemoptysis; had continuous anticoagulation treatment within 10 days before the study treatment;
5. Has experienced thromboembolic events such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism within 6 months before the study treatment;
6. Has active autoimmune or inflammatory diseases, or has a related history, including inflammatory bowel disease (such as colitis or Crohn's disease), diverticulitis (except diverticular disease), systemic lupus erythematosus, sarcoidosis syndrome or Wegener's syndrome (such as granulomatous vasculitis, Gray's disease, rheumatoid arthritis, pituitary inflammation and uveitis). There are the following exceptions: patients with vitiligo or alopecia; patients with stable hypothyroidism after hormone replacement therapy (such as after Hashimoto's thyroiditis); any patients with chronic skin diseases that do not require systemic treatment; patients who can be included within the past 5 years without active diseases, but only after consultation with the study doctor;
7. Active infections, including tuberculosis or human immunodeficiency virus (HIV 1/2 antibody positive);
8. Uncontrolled complications, including but not limited to: receiving study treatment for persistent or active infections (except HBV or HCV), symptomatic congestive heart failure, uncontrolled diabetes, uncontrolled hypertension, unstable angina pectoris, uncontrolled arrhythmia, active interstitial lung disease, severe chronic gastrointestinal diseases with diarrhea, or conditions that may limit compliance with study requirements, increase the risk of adverse events or affect the subject's ability to provide written informed consent;
9. Pregnant or lactating women;
10. The patient does not agree to use effective contraceptive measures during the treatment period and within the following 3 months;
11. Patients participating in other clinical studies simultaneously;
12. Patients with critical conditions unable to complete the survey;
13. Other primary malignant tumor history, but the following situations are excluded: malignant tumors treated for curative purposes, and having no known active diseases for ≥ 5 years before the study treatment and a low potential risk of recurrence; fully treated non-melanoma skin cancer or benign lentigo-like nevus without evidence of disease; fully treated carcinoma in situ with no evidence of disease;
14. Patients with a history of mental illness (such as schizophrenia, mania, anxiety disorder, depression, phobia, etc.) or patients diagnosed with mental illness during the clinical trial enrollment or their spouses;
15. Patients with communication disorders due to confusion, aphasia, or intellectual disability caused by reasons such as communication barriers or inability to answer normally;
16. Patients with other malignant tumor diseases;
17. Has a ≥ 3-grade allergy history to any component of vebecotota monoclonal antibody and/or pannipil monoclonal antibody injection and/or ivosizumab monoclonal antibody injection;
18. The investigator considers that there are other factors that are not suitable for inclusion or that may affect the subject's participation or completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
pCR | After surgery (approximately 9-10 weeks after start of study treatment)
  Pathological complete response rate

SECONDARY OUTCOMES:
MPR | After surgery (approximately 9-10 weeks after start of study treatment)
  major pathological remission

OTHER OUTCOMES:
ORR | 9-10 weeks
  objective response rate
EFS | 1 years
  event free survival
OS | 2 years
  overall survival

IPD SHARING:
Plan to Share IPD: Undecided